CLINICAL TRIAL: NCT04453839
Title: ZYESAMI (Aviptadil) Intermediate Population Expanded Access Protocol
Brief Title: ZYESAMI (Aviptadil) Intermediate Population Expanded Access Protocol (SAMICARE)
Acronym: SAMICARE
Status: No longer available | Type: Expanded Access
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Other Study IDs: ZYESAMI_EA-1
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-01

CONDITIONS: Critical COVID-19 With Respiratory Failure
MeSH Terms: interventions — aviptadil; Vasoactive Intestinal Peptide

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ZYESAMI (aviptadil acetate) — Patients will be treated with 12 hour infusions of ZYESAMI at ascending doses of 50/100/150 pmol/kg/hr on 3 or more successive days
  Other Names: Vasoactive Intestinal Peptide; VIP

SUMMARY:
Patients with Critical COVID-19 and respiratory failure who are ineligible for enrollment in NCT04311697, who live more than 50 miles from an existing collaborating research center, or who are already hospitalized and cannot safely be transferred to a collaborating research facility may be considered for expanded access by the sponsor.

Treating physicians must complete FDA Form 3396 and receive a letter of authorization from NeuroRx, along with local IRB authorization.

Please refer to FDA guidance for Individual Patient Expanded Access https://www.fda.gov/media/91160/download

DETAILED DESCRIPTION:
5. INTRODUCTION

5.1 Executive Summary ZYESAMI (aviptadil) is a synthetic form of Vasoactive Intestinal Polypeptide (VIP), a ubiquitous, naturally synthesized human peptide with extensively documented anti-inflammatory, anti-cytokine cascade properties. It has been granted FDA Fast Track Designation for treatment of Critical COVID-19 with Respiratory Failure. A phase 2/3 trial is underway that has passed its first evaluation at 30 patients for safety and futility. This expanded access protocol is designed to offer access to investigational use of RLF-100 to patients who do not qualify for inclusion in Protocol RLF-100-001 (NCT04311697) either on the basis of specific medical exclusions or because there is no accessible study site available to the prospective participant.

5.2 Definition of Critical COVID-19

In May 2020, FDA defined Critical COVID-19 to be used in clinical trials and disease staging as follows:

Critical COVID-19

* Positive testing by standard RT-PCR assay or an equivalent test
* Evidence of Respiratory Failure based on FDA definition of: need for Endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)

Acute Lung Injury in COVID-19 is characterized by progressive failure of corporeal oxygenation, attributed on large part by SARS-CoV-2 infection of Alveolar Type II cells (Mason 2020). Extensive nonclinical studies document that 70% of VIP in the body binds to receptors on the Alveolar Type II cell, where VIP is known to block cytokine production and upregulate production of surfactant.

Severity of COVID is associated with and graded by a progressively worsened state of oxygenation. This is seen in the PaO2/FIO2 ratio, which reflects the status of oxygenation for patients on high pressure oxygen and mechanical ventilation. In patients breathing room air, disease severity is assessed by SpO2. Many patients with Critical COVID meet the clinical definitions of Acute Respiratory Distress Syndrome (ARDS). However, there is increasing recognition that respiratory distress in COVID-19 has different characteristics than ARDS in the setting of bacterial sepsis and other common presentations of ARDS.

The pathologic hallmark of COVID-19 lung injury is diffuse alveolar damage, vascular endothelium damage, and damage to the surfactant-producing type II cells which results in loss of the integrity of the alveolar-capillary barrier, transudation of protein-rich fluid across the barrier, pulmonary edema, and hypoxemia from intrapulmonary shunting. Typically, patients who have progressed to Critical COVID-19 require care in an intensive care unit (ICU). The mortality rate is approximately 50%. Deaths usually result from multisystem organ failure rather than lung failure alone.

5.3 ZYESAMI Experimental Therapy in COVID-19

Under this protocol, patients with Critical COVID-19 will be treated with ZYESAMI (Aviptadil) with the aim to support pulmonary alveolar function, combat the cytokine-induced inflammation, improve blood oxygenation, and reduce mortality.

5.4 Clinical Rationale Given by intravenous infusion in appropriate concentrations, ZYESAMI has been shown in clinical trials to have a manageable safety profile with no observed SAEs to date that would rise to the level of a black box warning.

6. OBJECTIVES

6.1 Primary Objective The primary objective of this study is to measure the effectiveness and safety of ZYESAMI + maximal standard of care (SOC) in treating Critical COVID-19 with Respiratory Failure.

6.2 Secondary Objective The key secondary objective is to test the hypothesis that ZYESAMI improves blood oxygenation as measured by SaO2.

ELIGIBILITY:
Inclusion Criteria:

* Critical COVID-19 with Respiratory Failure

Exclusion Criteria:

* Patients who are eligible for enrollment in RLF-100_001 are excluded from this protocol and live within 50 miles of a study site for NCT04311697 cannot be enrolled unless already admitted to an ICU and ineligible for transfer
* Mean Arterial Pressure < 65 mm Hg with use of pressor per ICU protocol
* Irreversible condition (other than COVID-19) with projected fatal course
* ECMO
* Chemotherapy-induced neutropenia (granulocyte count <1000/mm3);
* Cardiogenic shock; congestive heart failure - NYHA Class 3 or 4;
* Liquid Diarrhea more than 3x/day; defined as more than 3 non-bloody watery stools within a 24-hour period, requiring additional fluid and electrolyte supplementation

Ages: 12 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Javitt, MD, MPH, Study Chair — NRx Pharmaceuticals, Inc.
Locations (25):
- United States (25):
  - Dignity Health-Mercy Gilbert Medical Center, Gilbert, Arizona
  - Honor Health Shea Medical Center, Scottsdale, Arizona
  - Kaiser Permanente, Baldwin Park, California
  - University of California - Irvine, Irvine, California
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Lakeland Regional Health, Lakeland, Florida
  - Miller School of Medicine / University of Miami Medical Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Baycare St. Joseph Hospital, Tampa, Florida
  - Southeast Georgia Health system, Brunswick, Georgia
  - Maui Health Systems, Wailuku, Hawaii
  - St. Anthony Regional Hospital, Carroll, Iowa
  - University of Louisville, Louisville, Kentucky
  - St. Tammany Parish Hospital, Covington, Louisiana
  - Our Ladies of Lourdes Regional Hospital, Lafayette, Louisiana
  - St. Joseph Heritage Healthcare, Saint Joseph, Missouri
  - Great Plains Health, North Platte, Nebraska
  - Self Regional Healthcare, Greenwood, South Carolina
  - Hendrick Medical Center, Abilene, Texas
  - Baptist Hospitals of Southeast Texas, Beaumont, Texas
  - Medical City Denton, Denton, Texas
  - HR Health Institute for Research & Development, Edinburg, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital Houston, Houston, Texas
  - Medical City McKinney, McKinney, Texas

REFERENCES:
- See also: Intravenous Aviptadil Is Associated with Increased Recovery and Survival in Patients with COVID-19 Respiratory Failure: Results of a 60-Day Randomized Controlled Trial — https://europepmc.org/article/ppr/ppr342295
- See also: Brief Report: Rapid Clinical Recovery From Critical Coronavirus Disease 2019 With Respiratory Failure in a Pregnant Patient Treated With IV Vasoactive Intestinal Peptide — https://journals.lww.com/ccejournal/Fulltext/2022/01000/Brief_Report__Rapid_Clinical_Recovery_From.1.aspx

DOCUMENTS (2):
  • Study Protocol (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04453839/Prot_001.pdf
  • Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04453839/ICF_002.pdf